CLINICAL TRIAL: NCT04403711
Title: The Effect of Adding Dexmedetomidine to the Local Anesthetic Solution for Ultrasonography-guided TAP Block in Inguinal Hernia Repair
Brief Title: Dexmedetomidine in TAP Block for Inguinal Hernia Repair
Acronym: TAP-dex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAP-dexmedetomidine
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Inguinal Hernia; Analgesia; Pain, Acute; Pain, Chronic; Pain, Neuropathic
Keywords: transversus abdominis plane block; dexmedetomidine
MeSH Terms: conditions — Hernia, Inguinal; Agnosia; Acute Pain; Chronic Pain; Neuralgia | interventions — Anesthetics, Local; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local anesthetic and dexmedetomidine (Active Comparator): ultrasound-guided transversus abdominis plane block with 25 mL ropivacaine 0.5% and 2 mL dexmedetomidine
  Interventions: Other: local anesthetic and dexmedetomidine
- local anesthetic and placebo (Placebo Comparator): ultrasound-guided transversus abdominis plane block with 25 mL ropivacaine 0.5% and 2 mL normal saline
  Interventions: Other: local anesthetic and placebo

INTERVENTIONS:
Other: local anesthetic and dexmedetomidine — in patients allocated to the dexmedetomidine group, ultrasound-guided transversus abdominis plane block will be performed with the combination of local anesthetic and dexmedetomidine
  Other Names: medication used in regional anesthetic technique
  Arms: local anesthetic and dexmedetomidine
Other: local anesthetic and placebo — in patients allocated to the dexmedetomidine group, ultrasound-guided transversus abdominis plane block will be performed with the combination of local anesthetic and normal saline
  Other Names: medication used in regional anesthetic technique
  Arms: local anesthetic and placebo

SUMMARY:
This prospective double-blind randomized study will aim at evaluating the short- and long-term postoperative analgesic efficacy of the ultrasound-guided transversus abdominis plane (TAP) block with a combination of local anesthetic and dexmedetomidine in inguinal hernia repair under general anesthesia

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most commonly performed surgical procedures worldwide, especially in the day-case setting. It can be accompanied by moderate to severe postoperative pain, which can delay return to normal daily activities or lead to the development of chronic pain. Chronic pain after hernia repair has a reported prevalence ranging between 0% and 43% with both nociceptive and neuropathic features. The transversus abdominis plane (TAP) block is an effective regional anesthetic technique to reduce postoperative pain intensity, time to first rescue anesthetic administration and opioid demand after upper and lower abdominal surgery. Dexmedetomidine is a selective α2-adrenergic agonist with analgesic properties that has been shown to prolong local anesthetic action when used as an adjunct to local anesthetic solutions in neuraxial anesthesia. The aim of this prospective, double-blind placebo controlled randomized study will be to evaluate the analgesic efficacy of ultrasound-guided TAP block where local anesthetic is supplemented by dexmedetomidine in patients undergoing unilateral elective inguinal hernia repair with the Lichtenstein technique under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) patients I-III undergoing inguinal hernia repair with a mesh
* open hernia repair
* elective surgery

Exclusion Criteria:

* inability to consent to the study due to language barriers or cognitive dysfunction -
* bilateral inguinal hernia repair,
* body mass index over 40 kg m-2,
* skin infection at the puncture site
* contraindication to paracetamol or non-steroidal anti-inflammatory drug (NSAIDs) administration
* known previous hepatic or renal impairment as assessed by the patients' history and routine biochemical markers
* coagulation abnormalities
* history of gastroesophageal reflux and preoperative use of opioids or NSAIDs for chronic pain conditions
* reoperation of recurrent inguinal hernia after previous mesh repair

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
pain score 3 hours postoperatively | 3 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 3 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

SECONDARY OUTCOMES:
incidence of chronic pain | 6 months after surgery
  occurrence of chronic pain at the site of the operation, with the use of the NRS, at rest and during movement

OTHER OUTCOMES:
morphine consumption | 24 hours postoperatively
  morphine consumption through patient-controlled analgesia device for 24 hours postoperatively
satisfaction from postoperative analgesia | 24 hours postoperatively
  satisfaction from postoperative analgesia on a four-point Likert scale with 1 marked as minimal satisfaction and 4 as maximal satisfaction
transversus abdominis plane-related complications | 48 hours postoperatively
  transversus abdominis plane-related complications at the site of the local anesthetic injection

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bay-Nielsen M, Perkins FM, Kehlet H; Danish Hernia Database. Pain and functional impairment 1 year after inguinal herniorrhaphy: a nationwide questionnaire study. Ann Surg. 2001 Jan;233(1):1-7. doi: 10.1097/00000658-200101000-00001. PMID 11141218
- [Background] Alfieri S, Amid PK, Campanelli G, Izard G, Kehlet H, Wijsmuller AR, Di Miceli D, Doglietto GB. International guidelines for prevention and management of post-operative chronic pain following inguinal hernia surgery. Hernia. 2011 Jun;15(3):239-49. doi: 10.1007/s10029-011-0798-9. Epub 2011 Mar 2. PMID 21365287
- [Background] Petersen PL, Mathiesen O, Torup H, Dahl JB. The transversus abdominis plane block: a valuable option for postoperative analgesia? A topical review. Acta Anaesthesiol Scand. 2010 May;54(5):529-35. doi: 10.1111/j.1399-6576.2010.02215.x. Epub 2010 Feb 17. PMID 20175754
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Mikkelsen T, Werner MU, Lassen B, Kehlet H. Pain and sensory dysfunction 6 to 12 months after inguinal herniotomy. Anesth Analg. 2004 Jul;99(1):146-151. doi: 10.1213/01.ANE.0000115147.14626.C5. PMID 15281521
- [Background] Goudarzi TH, Kamali A, Yazdi B, Broujerdi GN. Addition of dexmedetomidine, tramadol and neostigmine to lidocaine 1.5% increasing the duration of postoperative analgesia in the lower abdominal pain surgery among children: A double-blinded randomized clinical study. Med Gas Res. 2019 Jul-Sep;9(3):110-114. doi: 10.4103/2045-9912.266984. PMID 31552872
- [Background] Theodoraki K, Papacharalampous P, Tsaroucha A, Vezakis A, Argyra E. The effect of transversus abdominis plane block on acute and chronic pain after inguinal hernia repair. A randomized controlled trial. Int J Surg. 2019 Mar;63:63-70. doi: 10.1016/j.ijsu.2019.02.007. Epub 2019 Feb 12. PMID 30769214
- [Background] Chen Q, Liu X, Zhong X, Yang B. Addition of dexmedetomidine or fentanyl to ropivacaine for transversus abdominis plane block: evaluation of effect on postoperative pain and quality of recovery in gynecological surgery. J Pain Res. 2018 Nov 16;11:2897-2903. doi: 10.2147/JPR.S178516. eCollection 2018. PMID 30532583
- [Background] Ramya Parameswari A, Udayakumar P. Comparison of Efficacy of Bupivacaine with Dexmedetomidine Versus Bupivacaine Alone for Transversus Abdominis Plane Block for Post-operative Analgesia in Patients Undergoing Elective Caesarean Section. J Obstet Gynaecol India. 2018 Apr;68(2):98-103. doi: 10.1007/s13224-017-0990-7. Epub 2017 Apr 26. PMID 29662278